CLINICAL TRIAL: NCT00621777
Title: Extended Duration Pharmacotherapy for Prevention of Relapse to Smoking
Brief Title: A Study of Varenicline for Prevention of Relapse to Smoking in Patients With Schizophrenia or Bipolar Disorder
Acronym: SCRP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, A. Eden Evins, A. Eden Evins, MD, MPH, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC# 2007-P-002221; R01DA021245 (NIH)
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Smoking
Keywords: schizophrenia; bipolar disorder; varenicline; smoking cessation; relapse prevention; cognitive behavioral therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Smoking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Randomized Phase: Varenicline (Active Comparator): Varenicline is a partial agonist at alpha4beta2 nicotinic acetylcholine receptors (nAChRs) and a full agonist at alpha 7 nAChRs that has been shown to be effective for smoking cessation compared with placebo and bupropion, with effects on abstinence rates for up to one year. Varenicline has demonstrated safety when dosed at 1 mg twice per day for up to one year. Because varenicline, at a dose of 1 mg twice per day, may be a more effective treatment for sustained abstinence than bupropion, it was chosen as the medication intervention for this study.
  Interventions: Drug: Varenicline
- Randomized Phase: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — At each weekly study visit from the baseline visit to study week 11, ALL subjects will receive a one-week supply of varenicline with instructions on how to take the study medication. Titration is as follows: 0.5 mg varenicline per day for 3 days, then 0.5 mg twice per day for 4 days, and then 1 mg twice per day for 11 weeks.
  In addition, participants who enter the relapse prevention phase and are randomized to the varenicline condition will receive varenicline at the dose used to attain initial abstinence for 40 weeks.
  Other Names: Chantix
  Arms: Randomized Phase: Varenicline
Drug: Placebo — At each weekly study visit from the baseline visit to study week 11,ALL subjects will receive a one-week supply of varenicline with instructions on how to take the study medication. Titration is as follows: 0.5 mg varenicline per day for 3 days, then 0.5 mg twice per day for 4 days, and then 1 mg twice per day for 11 weeks.
  In addition, participants who enter the relapse prevention phase and are randomized to the placebo condition will receive placebo pills for 40 weeks.
  Arms: Randomized Phase: Placebo

SUMMARY:
Varenicline (Chantix) is a smoking cessation treatment that was approved in 2006 by the FDA for treatment of nicotine dependence and may be particularly beneficial in smokers with schizophrenia or bipolar disorder. Early experience with varenicline indicates that it will be effective for smoking cessation in schizophrenia and in addition, has the potential to be therapeutic for cognitive dysfunction in this population. In addition, more data is needed to evaluate the safety, tolerability and effectiveness of Varenicline in people with bipolar disorder.

To assess this possibility, we will evaluate the safety and efficacy of 12 months of varenicline in schizophrenia or bipolar disorder patients who are able to quit smoking in the short term with this treatment. To do so, we will enroll 324 smokers with schizophrenia or bipolar disorder from 6 mental health clinics in Massachusetts, New Hampshire, Michigan and Minnesota into an open, 12-week smoking cessation program that includes varenicline added to weekly group cognitive behavioral therapy (CBT). Those who achieve at least 2 weeks of continuous abstinence during the last 2 weeks of the open intervention will be randomized to the relapse prevention phase: a 40-week, double blind, placebo-controlled trial of varenicline at the dose used to quit smoking added to a tapering CBT schedule. Participants will then discontinue study medications and behavioral treatment and enter a 3-month follow up phase.

DETAILED DESCRIPTION:
Participants will be moderate to heavy smokers, aged 18-70, who have smoked an average of ≥10 cigarettes/day for the past year and who have not quit during the past year for a period >1 month.

During a 12-week open phase smoking cessation program, eligible subjects will be given active varenicline in addition to a 13-session weekly cognitive behavioral therapy program for smoking cessation. Dr. Evins (Principal Investigator) or a co-investigator will meet with subjects individually at Baseline of the Smoking Cessation Program to assess their medical eligibility for varenicline. A chart review will also be conducted by a research physician or psychiatrist.

Dr. Evins or another prescribing co-investigator will write a prescription for varenicline for each medically eligible subject. Subjects will receive their study medication at the end of each weekly group meeting. Any subject who experiences a serious side effect to the medication will meet with Dr. Evins or another medical co-investigator individually.

Subjects will set quit dates between the fourth and fifth CBT session weeks. Self-reports and exhaled carbon monoxide (CO) levels will be used to assess smoking status. Those subjects who have been abstinent for ≥2 weeks at the end of the 12th session group will be eligible for a 40-week relapse prevention program. After enrolling in the Relapse Prevention Program, subjects will be randomized to receive varenicline or placebos in addition to CBT for relapse prevention.

At Week 12 (the week before the end of the Smoking Cessation Program), Dr. Evins or another prescribing co-investigator will write prescriptions for subjects eligible for the randomized Relapse Prevention phase (i.e. successful quitters); these prescriptions will be sent to the Massachusetts General Hospital Research Pharmacy, where they will be filled according to the randomization code that the a research pharmacist will create.

When subjects come for the CBT orientation group session of the Relapse Prevention Program (Week 13), they will receive a 1-month supply of varenicline or placebo pill. During this randomized Relapse Prevention phase, medication compliance will be assessed at every group meeting by pill-count. Subjects will be asked about medication compliance and side effects at each group by the CBT group leaders and staff.

Any subject who experiences a serious side effect to the medication will meet with Dr. Evins or another medical co-investigator individually. In addition, Dr. Evins or a medical co-investigator will review the adverse events forms for each subject every week. Again, self-report and CO levels will be used to monitor smoking status.

Before and during both the open and randomized relapse prevention phases, subjects will be periodically assessed for cognitive performance, clinical characteristics, and adverse events in order to evaluate effects of withdrawal, predictors of cessation and relapse, and medication side effects. Following the completion of the 40-week relapse prevention phase, 3 follow-up assessments will be performed over a 3-month period to evaluate smoking status, cognitive functioning, and clinical effects.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18-70
* DSM-IV diagnosis of schizophrenia, schizoaffective disorder or bipolar disorder by diagnostic interview and chart review
* Smoke at least 10 cigarettes per day
* Clinically stable, on a stable dose of antipsychotic (schizophrenia) or mood stabilizer (bipolar) medication for at least 1 month
* No current active suicidal ideation
* Expired air carbon monoxide (CO) concentration >9 ppm
* Willing to take study medications and set a quit date within 2-3 weeks of beginning treatment and be willing to participate in the relapse prevention and follow-up portions of the study
* Women of childbearing potential must have a negative urine pregnancy test at baseline and agree to use an approved form of contraception during the study.

Exclusion Criteria:

* DSM-IV diagnosis of dementia, neurodegenerative disease, or other organic mental disorder
* Substance use disorder other than nicotine or caffeine in the last 6 months
* Major depressive disorder within the last 6 months
* Serious unstable medical illness including, cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease such that hospitalization for treatment of that illness is likely within the next 2 months
* Life-threatening arrhythmia or cerebro-vascular event within 6 months, cardiovascular event within 2 months or uncontrolled hypertension
* History of multiple head injuries with neurological sequelae, a single severe head injury with lasting neurological sequelae, or current CNS tumor
* Liver function tests elevated over twice normal
* Renal insufficiency with estimated creatinine clearance <40 ml/min
* Plan to continue use of tobacco products othe than cigarettes (e.g., cigar, pipe)
* Use of an investigational medication or device in the past 30 days
* Current suicidal or homicidal ideation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2008-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (10):
- United States (10):
  - University of Alabama Psychology Clinic, Birmingham, Alabama
  - Centerstone Research Institute, Bloomington, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts Mental Health Center, Boston, Massachusetts
  - Touchstone Innovare, Grand Rapids, Michigan
  - University of Minnesota Psychological Clinic, Minneapolis, Minnesota
  - West Central Behavioral Health, Claremont, New Hampshire
  - Riverbend Community Mental Health Center, Concord, New Hampshire
  - The Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - Community Council of Nashua, Nashua, New Hampshire

REFERENCES:
- [Background] From the Centers for Disease Control and Prevention. Annual smoking attributable mortality, years of potential life lost and economic costs--United States, 1995-1999. JAMA. 2002 May 8;287(18):2355-6. No abstract available. PMID 12001942
- [Background] Addington J, el-Guebaly N, Addington D, Hodgins D. Readiness to stop smoking in schizophrenia. Can J Psychiatry. 1997 Feb;42(1):49-52. doi: 10.1177/070674379704200107. PMID 9040923
- [Background] Adler LE, Olincy A, Waldo M, Harris JG, Griffith J, Stevens K, Flach K, Nagamoto H, Bickford P, Leonard S, Freedman R. Schizophrenia, sensory gating, and nicotinic receptors. Schizophr Bull. 1998;24(2):189-202. doi: 10.1093/oxfordjournals.schbul.a033320. PMID 9613620
- [Background] Barr, R.S.; Culhane, M.A.; Pizzagalli, D.; Goff, D.C.; and Evins, A.E. A double blind placebo controlled trial of the effects of transdermal nicotine on reward responsivity in non-smokers with schizophrenia. NIMH New Clinical Drug Evaluation Unit. Boca Raton, FL, 2006
- [Background] Breese CR, Lee MJ, Adams CE, Sullivan B, Logel J, Gillen KM, Marks MJ, Collins AC, Leonard S. Abnormal regulation of high affinity nicotinic receptors in subjects with schizophrenia. Neuropsychopharmacology. 2000 Oct;23(4):351-64. doi: 10.1016/S0893-133X(00)00121-4. PMID 10989262
- [Background] Carroll KM, Nich C, Sifry RL, Nuro KF, Frankforter TL, Ball SA, Fenton L, Rounsaville BJ. A general system for evaluating therapist adherence and competence in psychotherapy research in the addictions. Drug Alcohol Depend. 2000 Jan 1;57(3):225-38. doi: 10.1016/s0376-8716(99)00049-6. PMID 10661673
- [Background] de Leon J, Dadvand M, Canuso C, White AO, Stanilla JK, Simpson GM. Schizophrenia and smoking: an epidemiological survey in a state hospital. Am J Psychiatry. 1995 Mar;152(3):453-5. doi: 10.1176/ajp.152.3.453. PMID 7864277
- [Background] de Leon J, Diaz FJ, Rogers T, Browne D, Dinsmore L. Initiation of daily smoking and nicotine dependence in schizophrenia and mood disorders. Schizophr Res. 2002 Jul 1;56(1-2):47-54. doi: 10.1016/s0920-9964(01)00217-1. PMID 12084419
- [Background] Evins AE, Cather C, Rigotti NA, Freudenreich O, Henderson DC, Olm-Shipman CM, Goff DC. Two-year follow-up of a smoking cessation trial in patients with schizophrenia: increased rates of smoking cessation and reduction. J Clin Psychiatry. 2004 Mar;65(3):307-11; quiz 452-3. doi: 10.4088/jcp.v65n0304. PMID 15096068
- [Background] Evins AE, Cather C, Deckersbach T, Freudenreich O, Culhane MA, Olm-Shipman CM, Henderson DC, Schoenfeld DA, Goff DC, Rigotti NA. A double-blind placebo-controlled trial of bupropion sustained-release for smoking cessation in schizophrenia. J Clin Psychopharmacol. 2005 Jun;25(3):218-25. doi: 10.1097/01.jcp.0000162802.54076.18. PMID 15876899
- [Background] Gonzales D, Rennard SI, Nides M, Oncken C, Azoulay S, Billing CB, Watsky EJ, Gong J, Williams KE, Reeves KR; Varenicline Phase 3 Study Group. Varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs sustained-release bupropion and placebo for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):47-55. doi: 10.1001/jama.296.1.47. PMID 16820546
- [Background] Hughes JR, Hatsukami DK, Mitchell JE, Dahlgren LA. Prevalence of smoking among psychiatric outpatients. Am J Psychiatry. 1986 Aug;143(8):993-7. doi: 10.1176/ajp.143.8.993. PMID 3487983
- [Background] Jorenby DE, Hays JT, Rigotti NA, Azoulay S, Watsky EJ, Williams KE, Billing CB, Gong J, Reeves KR; Varenicline Phase 3 Study Group. Efficacy of varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs placebo or sustained-release bupropion for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):56-63. doi: 10.1001/jama.296.1.56. PMID 16820547
- [Background] Mihalak KB, Carroll FI, Luetje CW. Varenicline is a partial agonist at alpha4beta2 and a full agonist at alpha7 neuronal nicotinic receptors. Mol Pharmacol. 2006 Sep;70(3):801-5. doi: 10.1124/mol.106.025130. Epub 2006 Jun 9. PMID 16766716
- [Background] Diaz FJ, James D, Botts S, Maw L, Susce MT, de Leon J. Tobacco smoking behaviors in bipolar disorder: a comparison of the general population, schizophrenia, and major depression. Bipolar Disord. 2009 Mar;11(2):154-65. doi: 10.1111/j.1399-5618.2009.00664.x. PMID 19267698
- [Derived] Cather C, Hoeppner S, Pachas G, Pratt S, Achtyes E, Cieslak KM, Evins AE. Improved Depressive Symptoms in Adults with Schizophrenia During a Smoking Cessation Attempt with Varenicline and Behavioral Therapy. J Dual Diagn. 2017 Jul-Sep;13(3):168-178. doi: 10.1080/15504263.2017.1319585. Epub 2017 Apr 17. PMID 28414583
- [Derived] Thorndike AN, Achtyes ED, Cather C, Pratt S, Pachas GN, Hoeppner SS, Evins AE. Weight gain and 10-year cardiovascular risk with sustained tobacco abstinence in smokers with serious mental illness: a subgroup analysis of a randomized trial. J Clin Psychiatry. 2016 Mar;77(3):e320-6. doi: 10.4088/JCP.15m10074. PMID 27046320
- [Derived] Evins AE, Cather C, Pratt SA, Pachas GN, Hoeppner SS, Goff DC, Achtyes ED, Ayer D, Schoenfeld DA. Maintenance treatment with varenicline for smoking cessation in patients with schizophrenia and bipolar disorder: a randomized clinical trial. JAMA. 2014 Jan 8;311(2):145-54. doi: 10.1001/jama.2013.285113. PMID 24399553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled from 03/08 to 04/12 from 10 community mental health centers in MA, MI, NH, IN, AL, and MN, participants were 18-70 years, outpatients with schizophrenia, schizoaffective or bipolar disorder, smoked 10+ cigs/day, had CO levels >9 ppm, willing to take varenicline, agreed to set a quit date within 4 wks of enrollment, and were stable
Pre-assignment Details: 44 participants were excluded after signing consent: 4 site closure, 40 Did not meet inclusion criteria, 17 Active substance abuse, 8 Unstable medical condition, 8 Unstable psychological symptoms, 4 Lost to follow-up, 3 Other
Groups:
- Varenicline: Varenicline is a partial agonist at alpha4beta2 nicotinic acetylcholine receptors (nAChRs) and a full agonist at alpha 7 nAChRs that has been shown to be effective for smoking cessation compared with placebo and bupropion, with effects on abstinence rates for up to one year.
  1. Open label, smoking cessation phase: At each weekly study visit from the baseline visit to study wk 11, ALL subjects will receive a one-week supply of varenicline as follows: 0.5 mg varenicline per day for 3 days, then 0.5 mg twice per day for 4 days, and then 1 mg twice per day for 11 wks.
  2. Double-Blind, Placebo-Controlled, Relapse-Prevention Phase:
  Participants in the open phase who met criteria for biochemically verified, 7-day, point-prevalence abstinence at wks 11 and 12 were considered to be continuously abstinent for at least 14 days and were randomized to continue varenicline, 1.0 mg twice a day, or switch to identical-appearing placebo for wks 12 through 52
Period: Open Phase
Arm/Group | Varenicline | Placebo
Started | 203 | 0 (During this open label phase, all study participants received varenicline)
Completed | 87 | 0
Not Completed | 116 | 0
Not completed — Adverse Event | 20 | 0
Not completed — Did not abstain during open phase | 56 | 0
Not completed — Withdrawal by Subject | 17 | 0
Not completed — administrative | 13 | 0
Not completed — Lost to Follow-up | 10 | 0
Period: Randomized Phase
Arm/Group | Varenicline | Placebo
Started | 40 (87 open phase participants were continuously abstinent for at least 14 days and were randomized) | 47
Completed | 33 | 28
Not Completed | 7 | 19
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 1 | 9
Not completed — administrative | 0 | 3
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Varenicline: Varenicline is a partial agonist at alpha4beta2 nicotinic acetylcholine receptors (nAChRs) and a full agonist at alpha 7 nAChRs that has been shown to be effective for smoking cessation compared with placebo and bupropion, with effects on abstinence rates for up to one year. Varenicline has demonstrated safety when dosed at 1 mg twice per day for up to one year.
  Varenicline: At each weekly study visit from the baseline visit to study week 11, ALL subjects will receive a one-week supply of varenicline with instructions on how to take the study medication. Titration is as follows: 0.5 mg varenicline per day for 3 days, then 0.5 mg twice per day for 4 days, and then 1 mg twice per day for 11 weeks.
  In addition, participants who enter the relapse prevention phase and are randomized to the varenicline condition will receive varenicline at the dose used to attain initial abstinence for 40 weeks.
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 40 | 47 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (9.6) | 45.7 (10.3) | 47.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 24 | 31 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 30 | 34 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 7 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 38 | 47 | 85
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of 7-day Point Prevalence Abstinence at the End of the Relapse Prevention Phase (Study Week 53) in the Extended Duration Pharmacotherapy Group vs. the Placebo Group
Time Frame: 76 weeks
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 40 | 47
participants
  7-day, point-prevalence abstinence at week 52 | 24 | 9
  Continuous abstinence, weeks 12-64 | 18 | 7
  Continuous abstinence, weeks 12-76 | 12 | 5

2. Secondary Outcome: Safety and Tolerability of Extended Duration Pharmacotherapy When Added to Antipsychotic Medications in Schizophrenia Patients Who Have Recently Quit Smoking as Assessed by the Brief Psychiatric Rating Scale
Description: Brief Psychiatric Rating Scale is a 24 item scale that is designed to assess positive and negative symptoms, and general psychopathology in people with serious mental illness. Each item is rated on a 7-point scale from not present to extremely severe; higher scores in a range of 24 to 168, indicate more severe symptoms Ratings are based on observation and patient report. The validity of the BPRS is generally high when compared with other measures of general psychopathology. It was administered at baseline, study weeks 12, 18, 26, 38, 52
Time Frame: at week 52
Population: Only 63 subjects completed study visit #52, therefore only these subjects were analyzed at this time point for this variable
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 31 | 32
units on a scale | 50.43 (15.08) | 47.88 (12.12)

3. Secondary Outcome: Effect of Treatment With Varenicline Versus Placebo on Health-related Quality of Life Indices in Recently Abstinent Smokers With Schizophrenia or Bipolar Disorder as Measured by the 12-Item Short Form Health Survey (SF-12)
Description: The 12-Item Short Form Health Survey (SF-12) is a 12-item measure of perceived health status with good reliability, validity and correlation with other health measures. It is scored via a standard algorithm, with higher scores indicating better patient self perception of health, with a mean score of 50 and a standard deviation of 10 in a representative sample of the US population. The score is computed using the scores of the twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health. This was administered at baseline and end of study.
Time Frame: at week 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 47.59 (10.95) | 48.39 (9.05)

ADVERSE EVENTS:
Time Frame: At every visit: Calgary Depression Scale, the Montgomery-Asberg Depression and the Young Mania Rating Scales. AEs were ascertained by general/specific query: headache, nausea, vomiting, tachycardia, excitement, agitation, anxiety, insomnia, irritability.
Description: Additional assessments were conducted at baseline; at study weeks 12, 18, 26, 38, 52, and 64; the Brief Psychiatric Rating Scale, Schedule for the Assessment of Negative Symptoms and assessments for health-related quality of life were conducted at baseline and weeks 12, 52, and 64.
Groups:
- Varenicline Open Label (Open Phase): Varenicline is a partial agonist at alpha4beta2 nicotinic acetylcholine receptors (nAChRs) and a full agonist at alpha 7 nAChRs that has been shown to be effective for smoking cessation compared with placebo and bupropion, with effects on abstinence rates for up to one year.
  1. Open label, smoking cessation phase: At each weekly study visit from the baseline visit to study wk 11, ALL subjects will receive a one-week supply of varenicline as follows: 0.5 mg varenicline per day for 3 days, then 0.5 mg twice per day for 4 days, and then 1 mg twice per day for 11 wks.
- Varenicline: Varenicline is a partial agonist at alpha4beta2 nicotinic acetylcholine receptors (nAChRs) and a full agonist at alpha 7 nAChRs that has been shown to be effective for smoking cessation compared with placebo and bupropion, with effects on abstinence rates for up to one year.
  2. Double-Blind, Placebo-Controlled, Relapse-Prevention Phase: Participants in the open phase who met criteria for biochemically verified, 7-day, point-prevalence abstinence at wks 11 and 12 were considered to be continuously abstinent for at least 14 days and were randomized to continue varenicline, 1.0 mg twice a day, or switch to identical-appearing placebo for wks 12 through 52
- Placebo: 2. Double-Blind, Placebo-Controlled, Relapse-Prevention Phase: Participants in the open phase who met criteria for biochemically verified, 7-day, point-prevalence abstinence at wks 11 and 12 were considered to be continuously abstinent for at least 14 days and were randomized to continue varenicline, 1.0 mg twice a day, or switch to identical-appearing placebo for wks 12 through 52
Arm/Group | Varenicline Open Label (Open Phase) | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 3/203 | 4/40 | 7/47
Other Adverse Events (participants affected / at risk) | 113/203 | 26/40 | 21/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline Open Label (Open Phase) (N=203) | Varenicline (N=40) | Placebo (N=47)
Sepsis associated with complications of diabetes that resulted in death (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — medical hospitalization
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — medical hospitalization
Pancreatitis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — medical hospitalization
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — medical hospitalization
psychiatric hospitalization (Psychiatric disorders) | 3 (3) | 2 (2) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline Open Label (Open Phase) (N=203) | Varenicline (N=40) | Placebo (N=47)
Nausea (General disorders) | 113 (340) | 25 (69) | 18 (52)
Anxiety (Psychiatric disorders) | 88 (266) | 19 (81) | 19 (53)
Irritability (Psychiatric disorders) | 83 (204) | 14 (58) | 18 (47)
Headache (General disorders) | 86 (222) | 26 (66) | 21 (64)
Agitation (Psychiatric disorders) | 88 (189) | 18 (56) | 19 (53)
Excitement (Psychiatric disorders) | 85 (172) | 17 (49) | 21 (44)
Insomnia (General disorders) | 81 (237) | 21 (82) | 21 (67)
Vomiting (Gastrointestinal disorders) | 71 (137) | 17 (48) | 12 (22)
Tachycardia (Cardiac disorders) | 39 (89) | 10 (19) | 16 (29)
Abnormal dreams (General disorders) | 36 (119) | 8 (44) | 11 (45)
Chest pain (Cardiac disorders) | 8 (13) | 4 (11) | 2 (9)
Constipation (Gastrointestinal disorders) | 14 (38) | 3 (8) | 3 (16)
Lightheaded (General disorders) | 21 (45) | 5 (31) | 4 (12)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (12) | 6 (11) | 2 (7)
Fatigue (General disorders) | 7 (20) | 3 (14) | 2 (5)
Suicidal Ideation (Psychiatric disorders) | 6 (6) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No